CLINICAL TRIAL: NCT05645094
Title: Neoadjuvant Envafolimab in Resectable and Locally Advanced MSI-H/dMMR Rectal Cancer: a Single-arm, Prospective Trial
Brief Title: Neoadjuvant Envafolimab in Resectable and Locally Advanced MSI-H/dMMR Rectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, LI XIN-XIANG, Professor, Fudan University
Other Study IDs: FDCRC85LXX
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Locally Advanced Rectal Carcinoma; MSI-High
MeSH Terms: interventions — envafolimab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Envafolimab — Patients will receive single drug therapy of Envafolimab (300mg) once every two weeks. Patients who do not have tumor regression after 3 months of treatment should be judged by the investigator whether to adopt standard chemoradiotherapy plus surgery. Patients with tumor regression should continue to receive Envafolimab therapy until 6 months. For patients who do not reach complete clinical response (cCR) after 6 months of treatment, the investigator shall determine whether to perform standard chemoradiotherapy or radical surgery. For patients who reach cCR, they could receive the observation waiting or local resection which depend on the investigator. Patients should be followed up until reaching cCR or 3 years after surgery.

SUMMARY:
This is a single center, prospective, single arm clinical trial to evaluate the efficacy and safety of Envafolimab as a neoadjuvant therapy for resectable and locally advanced dMMR or MSI-H rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects volunteer to join the study and could complete the signing of the informed consent form, and had good compliance;
2. Age ≥ 18 years old and<80 years old (when signing the informed consent form);
3. ECOG score 0-1;
4. Resectable rectal cancer was confirmed by pathological diagnosis (pathology/cytology) and imaging;
5. The clinical TNM stage is T3-4N0M0 or TanyN+M0;
6. The distance from the lower edge of the tumor to the lower edge of the anus is ≤ 10cm;
7. Patients who need routine neoadjuvant therapy after evaluation;
8. dMMR or MSI-H was detected by immunohistochemistry/PCR;
9. Patients did not received immunotherapy, chemotherapy, targeted therapy or radiotherapy for rectal cancer in the past;
10. The expected life span exceeds 3 months;
11. It has measurable lesions (according to iRECIST standard, the long diameter of CT scan for non lymph node lesions is ≥ 10 mm, and the short diameter of CT scan for lymph node lesions is ≥ 15 mm);
12. The function of main organs is normal, they should meet the following standards:

    1. Blood routine examination: Absolute Neutrophil Count (ANC) 1.5 × 109/L, Platelet (PLT) ≥ 70 × 109/L, Hemoglobin (HGB) ≥ 90 g/L;
    2. Liver function: total bilirubin (TBIL) ≤ 1.5 × Upper Limit of Normal Value (ULN); Alanine Aminotransferase (ALT) and Aspartate Transferase (AST) ≤ 3 × ULN; Serum albumin ≥ 28 g/L; Alkaline phosphatase (ALP) ≤ 5 × ULN; After routine liver protection treatment, it meets the above criteria, and can be stable for at least 1 week. After evaluation by the researcher, it can be included in the group;
    3. Renal function: serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/mi (using the standard Cockcroft Gault formula);
    4. Coagulation function: International Normalized Ratio (INR) ≤ 1.5/PT ≤ 1.5 × ULN，aPTT≤1.5 × ULN; If the subject is receiving anticoagulation treatment, PT and INR should be within the scope of anticoagulation drugs.
    5. Thyroid function: normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is beyond the normal range, the subjects whose total T3 (or FT3) and FT4 are within the normal range can also be included in the group;
13. Female patients must be non pregnant and non lactating, and need to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill or condom) during the study treatment period and at least 120 days after the end of the study. During this period, it is not allowed to donate eggs to others or freeze them for fertilization and reproduction.

Exclusion Criteria:

1. Patients with active autoimmune diseases or autoimmune diseases that may recur are as follows, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, and those who have previously undergone thyroid surgery cannot be included; Subjects who suffer from vitiligo or asthma in childhood has completely alleviated, and do not need any intervention after adulthood can be included; Asthma requiring medical intervention with bronchodilators was excluded;
2. Subjects with any severe and/or uncontrollable disease. include:

   1. Poor blood pressure control (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg);
   2. Suffering from ≥ grade 2 myocardial ischemia or myocardial infarction, arrhythmia (QTc ≥ 470ms) and ≥ grade 2 congestive heart failure (NYHA classification);
   3. Active or uncontrolled serious infection (≥ CTCAE level 2 infection) requiring systemic anti bacterial, anti fungal or anti-virus treatment, including tuberculosis infection. Active hepatitis (transaminase does not meet the inclusion criteria, hepatitis B reference: HBV DNA ≥ 2000 IU/ml or ≥ 104 copies/ml; hepatitis C reference: HCV RNA ≥ 2000 IU/ml or ≥ 104 copies/ml; after nucleotide antiviral treatment, it is lower than the above criteria, it can be included in the group); Chronic hepatitis B virus carriers, HBV DNA<2000 IU/ml, must receive antiviral treatment at the same time during the trial to be included in the group;
   4. Renal failure requiring hemodialysis or peritoneal dialysis;
   5. Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
3. Poor control of diabetes (fasting blood glucose [FBG]>10mmol/L);
4. Those who received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before the start of the study treatment; Or there is a wound or fracture that has not been cured for a long time;
5. Serious arteriovenous thrombotic events occurred within 6 months before the study treatment, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
6. Those who have a history of abuse of psychotropic substances and are unable to quit or have mental disorders;
7. Tumor related symptoms and treatment:

   1. Within 3 weeks before the start of the study treatment, he had received surgery, chemotherapy, small molecule targeted therapy, radiotherapy or other anti-tumor therapy (washout period is calculated from the end time of the last treatment).
   2. Within 2 weeks before the start of the study, those who have received the treatment of Chinese patent drugs with anti-tumor indications specified in the NMPA approved drug manual (including compound cantharis capsule, Kangai injection, Kanglaite capsule/injection, Aidi injection, Brucea javanica oil injection/capsule, Xiaoaiping tablet/injection, cinobufagin capsule, etc.);
   3. Uncontrolled pleural effusion, pericardial effusion or ascites that still need repeated drainage (judged by the investigator);
8. Study treatment related:

   1. The history of live attenuated vaccine vaccination within 14 days before the start of the study treatment or the plan for live attenuated vaccine vaccination during the study period;
   2. Severe hypersensitivity reaction occurred after using monoclonal antibody;
   3. Active autoimmune diseases requiring systemic treatment (such as the use of disease relieving drugs, corticosteroids or immunosuppressants) occurred within 2 years before the start of the study treatment, except for substitution therapy (such as thyroxine, insulin or physiological corticosteroids for adrenal or pituitary insufficiency);
   4. Diagnosed as immune deficiency or being treated with systemic glucocorticoid or any other form of immunosuppressive therapy. (dosage>10mg/day prednisone or other effective hormones), and continue to use within 2 weeks after the first administration;
   5. Have a history of active tuberculosis;
9. Those who are participating in or have participated in other clinical researches within 4 weeks before the start of the study;
10. Have a history of severe allergy;
11. Known allergy to the active ingredient or excipient of Envafolimab;
12. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the subject or affect the completion of the study, or subjects who believe that there are other reasons that are not suitable for inclusion.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Resectable locally advanced dMMR or MSI-H rectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
cCR and pCR rates | 1-year
  Complete clinical response rate (cCR) after neoadjuvant therapy or complete pathological response rate (pCR) of patients undergoing surgery

SECONDARY OUTCOMES:
Tumor regression grade (TRG) | 1-year
  Surgical excision specimens are taken every 1 cm, and the sections are given to at least 2 pathologists for independent scoring
Objective response rate (ORR) | 1-year
local regrowth rate after cCR | 3-year
3-year relapse-free survival | 3-year
  relapse-free survival refers to the period of time between the date of surgery and the day of the patient's tumor recurrence or death (earliest occurrence).
3-year overall survival | 3-year
  For patients who still survive when the final analysis takes place, the date of the last 1 contact will be recorded.
Patients' quality of life | 3-month, 6-month, 9-month, 12-month, 18-month, 24-month
  The European Organization for Research and Treatment (EORTC)-QLQ-C30 HRQL questionnaire was assessed with repeated measures at regular intervals postoperatively at months 3, 6, 9, 12, 18, and 24
Acute toxicity associated with Envafolimab | from the beginning of treatment to 90 days after the end of Envafolimab
  According to the NCI CTCAE v5.0 assessment, the proportion of patients with treatment-related acute toxicity developed from the beginning of treatment to 90 days after the end of Envafolimab

CONTACTS AND LOCATIONS:
Overall Officials: Xinxiang Li, MD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No